CLINICAL TRIAL: NCT01603927
Title: Detect InSpect ChAracterise Resect and Discard 2
Acronym: DISCARD2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: University of Durham (Other)
Responsible Party: Sponsor
Other Study IDs: DISCARD2; PB-PG-1010-23222 (Other Grant/Funding Number: NHS National Institute for Health Research)
Record Dates: First submitted 2012-05-17; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colonoscopy with Narrow band imaging (NBI): All patients attending for routine colonoscopies performed for the diagnosis of symptoms or asymptomatic screening.
  Interventions: Device: Narrow band imaging for 'optical diagnosis' of colonic polyps (Olympus).

INTERVENTIONS:
Device: Narrow band imaging for 'optical diagnosis' of colonic polyps (Olympus). — Colonoscopists will narrow band imaging to provide an 'optical diagnosis' for colonic polyps found during routine colonoscopies performed for the diagnosis of symptoms or asymptomatic screening.

SUMMARY:
Bowel cancer is a common disorder in the UK. Most cancers happen when a type of polyp, called an adenoma, becomes cancerous. Polyps are growths in the large bowel that can be cancerous, non-cancerous, or pre-cancerous (adenoma). Polyps are most commonly detected during colonoscopy (camera test of the lower bowel). The removal of adenomas has been shown to reduce the subsequent risk of bowel cancer. Current practice is that all polyps are removed or biopsied to allow a laboratory diagnosis (histology). This is important as it influences if and when patients require follow-up colonoscopies, known as the surveillance interval. Patients with only non-cancerous polyps do not need surveillance.

A new blue light technology, called narrow band imaging (NBI), used during colonoscopy can help colonoscopists (doctor or nurse performing the procedure)differentiate between polyp types during colonoscopy. NBI is currently available in a large number of UK endoscopy units however is variably used. Studies from 'expert' centres have demonstrated that NBI allows accurate optical diagnosis of colonic polyps. Benefits of optical diagnosis include avoiding removal of non-cancerous polyps and an immediate (on the day) diagnosis for the patient including the surveillance interval.

The primary aim of this study is to evaluate the accuracy with which colonoscopists assess the required surveillance interval using optical diagnosis when compared with histology in non-expert centres. The investigators will invite 2500 patients, who have been referred for colonoscopy, to participate. Patients will undergo a routine colonoscopy the only addition being the use of NBI during the procedure. Colonoscopists will provide an optical diagnosis at the time of colonoscopy in addition to polyp removal or biopsy.

The investigators will compare surveillance intervals provided using optical diagnosis with the diagnosis from histology and thereby the accuracy with which colonoscopists can use the technology. The investigators will also calculate the cost savings to the NHS.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) continues to be a major problem in the UK and is the second most common cause of cancer death. The annual incidence is approximately 30,000 cases with an annual mortality rate of in the region of 16,000 (1). Most sporadic non-hereditary CRCs arise from benign colorectal adenomas (2). The detection and resection of colorectal adenomas at colonoscopy has been shown to reduce the subsequent risk of CRC by as much as 80% (3).

The NHS Bowel Cancer Screening Programme (BCSP) began roll-out in 2006 in England and as of April 2010, was established across 99.4% of the country. The BCSP is based on a strategy of biennial faecal occult blood test (FOBt) screening for men and women aged 60-75, followed by colonoscopy for those who test positive. Among its aims is the detection and resection of potentially pre-malignant colorectal adenomas thereby potentially reducing the incidence of CRC. The introduction of the BCSP has resulted in a dramatically increased demand for colonoscopy. To date approximately 80,000 colonoscopies have been performed within the BCSP and at least one adenoma found in just under half of the procedures (4). In addition, from 2012, the BCSP will introduce flexible sigmoidoscopy screening for all individuals aged 55 yr olds. This extrapolates to approximately 500,000 flexible sigmoidoscopies per year, with at least one polyp expected to be found in 75,000 procedures.

Greater than 90% of polyps detected at colonoscopy are small (6-9mm) or diminutive (≤5mm), with the latter making up the majority (5-7). In addition, approximately 50% of small polyps are non-neoplastic (8), known as adenomas. The number of adenomas present strongly influences the future risk of the development of advance neoplasia for the individual patient and therefore determines decisions on future surveillance intervals. As a result even small polyps, with little risk of harbouring cancer, are currently sent for histological assessment in order to determine whether or not they are adenomatous (9-11).

The ability to correctly diagnose a small polyp (< 10mm) during colonoscopy as adenomatous or non-adenomatous from its endoscopic characteristics (optical diagnosis) would allow small adenomas to be resected and discarded without the need to retrieve the polyp for formal histological assessment. Additionally, hyperplastic rectosigmoid polyps can be left in situ thereby reducing the need for polypectomy and the associated risks. Optical diagnosis would also enable surveillance intervals to be determined immediately after colonoscopy thereby avoiding the need for out-patient follow up, potentially leading to significant time and cost savings. Notably, histological assessment is an imperfect current gold standard as polyps may be lost or be unable to be assessed due to diathermy artefact in 8-25% of cases. Furthermore, standard histological techniques may misclassify up to 15% of adenomas as benign lesions.

Narrow band imaging (NBI; Olympus, Japan (12, 13)) is a new 'blue light' optical imaging modality available at a push of a button on the colonoscope head. By enhancing mucosal detail and in particular vascular structures it allows assessment of microvascular density (vascular pattern intensity - VPI (14); meshed brown capillary network (15-17)). Neoplastic tissue is characterized by increased angiogenesis and, therefore, adenomas appear darker when viewed with NBI. The use of microvascular assessment appears to have a short learning curve, as short as 60 histologically verified polyps (18-20), making it a potentially attractive and practical option for optical diagnosis. There are no known adverse events associated with NBI.

Two studies to date have assessed clinical implications of endoscopic diagnosis of small polyps on surveillance intervals using white light in combination with NBI. A study of diminutive polyps (≤5 mm) performed by a single expert colonoscopist (21), 134 out of 136 (98.5%) of patients would have had the same surveillance intervals when recommendations based on optical and histological diagnoses were compared. Similar results were reported in a study performed by three of the co-applicants (AI, JEE, BPS)(22) where 82 out of 130 patients could be given a surveillance interval immediately after colonoscopy based on optical diagnosis alone and the same interval was found after formal histopathology in 80 patients (98%) using British Society of Gastroenterology guidelines (23). Optical diagnosis accurately diagnosed 186 of 198 adenomas (sensitivity 0.94; 95% CI 0.90-0.97) and 55 of 62 hyperplastic polyps (specificity 0.89; 0.78 -0.95) with an overall accuracy of 241 of 260 (0.93; 0.89-0.96) for small polyp characterisation. In this study, using simple cost analysis, the authors estimated that optical diagnosis would have resulted in 77% cost savings for polyp analysis and clinical follow up (£13343 for 130 patients examined). Using Markov modelling, Hassan et al modelled the cost-effectiveness of 'resect and discard policy' and found that using it for diminutive polyps (≤5mm) would result in annual saving of $33 million when applied to colonoscopy screening of the US population (corresponding to overall saving of $330 million, assuming cumulative period of 10 years to screen just under a quarter of US population) (24).

Optical diagnosis may therefore benefit:

1. Patients: Shorter, more accurate examinations with fewer complications as a results of fewer polypectomies (less perforation and bleeding), reduced anxiety (awaiting histology results) and more appropriate use of endoscopic surveillance programmes.
2. NHS and other Healthcare providers: Increased efficiency (shorter lists, more exams per endoscopy list, fewer out-patient appointments, avoids unnecessary use of histology capacity) and reduced risk (fewer complications and fewer polyp 'misses'). Since the need for histology is set to greatly increase with an expansion of screening, a move to the routine use of NBI may substantially reduce the need to expand histology services.

We foresee no significant constraints to adoption of optical diagnosis as financial costs should be easily offset by savings from the efficiency benefits described above as 90% of polyps detected at colonoscopy are <10mm in size and therefore suitable for optical biopsy.

Study Design DISCARD 2 is a blinded calibration diagnostic study which will compare NBI optical diagnosis with histological assessment (as a reference standard) for patients with small polyps (<10mm) identified at colonoscopy

Recruitment Patients who are due to attend for a routine colonoscopy will be identified during out-patient clinics, during colonoscopy booking, or on the day of colonoscopy at each of the participating sites. Patients will be sent or given an information pack containing an information sheet and consent form. There will be two phases of recruitment to the study. All consenting patients undergoing colonoscopy are included in phase 1 of the study. Those who undergo a complete colonoscopy and in whom one or polyp <10mm in diameter is found will enter phase 2 of the study.

More detail regarding inclusion and exclusion criteria and outcome measures are provided below.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

1. Patients able to provide valid informed consent.
2. Patients over 18 years of age.
3. Patients attending for routine colonoscopy.

Phase 2

1. Patient fulfils inclusion criteria for phase 1.
2. Patients with one or more polyps under 10mm detected at colonoscopy.
3. Patients undergoing a complete colonoscopy confirmed by photo documentation of caecal landmarks.

Exclusion Criteria:

1. Patients with known inflammatory bowel disease (ulcerative colitis of Crohns disease) or known polyposis syndromes.
2. Patients who lack capacity to give informed consent as assessed by the clinical study team member taking consent.
3. Patients who are known to be pregnant (self-reported).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending for routine diagnostic or screening colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity NBI optical diagnosis in determining colonoscopy surveillance intervals. | 12 months
  The proportion of individuals requiring surveillance colonoscopy (according to British Society of Gastroenterology Guidelines)that are correctly identified by NBI optical diagnosis (test sensitivity).

SECONDARY OUTCOMES:
The sensitivity, specificity and accuracy of optical diagnosis on a per polyp basis. | 12 months
  Sensitivity, specificity and accuracy of optical diagnosis on a per-polyp basis
The learning curve and maintenance of accuracy of optical diagnosis. | 12 months
  Learning curve and maintenance of quality of optical diagnosis measured by proportion of polyps/patients diagnosed with high/low confidence.
The economic implications of replacing histological assessment with optical diagnosis. | 12 months
  Potential cost saving of optical diagnosis
Description of the population undergoing routine colonoscopy and prevalence of polyps and polyp type. | 12 months
  Proportion of patients with no polyps, small polyps, large polyps, categorised by age, gender and polyps type.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - County Durham and Darlington NHS Foundation Trust, Darlington, County Durham
  - North Cumbria University Hospitals NHS Trust, Carlisle, Cumbria
  - Northumbria Healthcare NHS Trust, Ashington, Northumberland
  - South Tees NHS Trust, Middlesbrough, Teeside
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees, Teeside

REFERENCES:
- [Background] National Bowel Cancer Audit 2009 NBOCAP Available at: http://www.nbocap.org.uk/resources/reports/NBOCAP_2009.pdf
- [Background] Morson B. President's address. The polyp-cancer sequence in the large bowel. Proc R Soc Med. 1974 Jun;67(6 Pt 1):451-7. doi: 10.1177/00359157740676P115. No abstract available. PMID 4853754
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Lee TJ, Rutter MD, Blanks RG, Moss SM, Goddard AF, Chilton A, Nickerson C, McNally RJ, Patnick J, Rees CJ. Colonoscopy quality measures: experience from the NHS Bowel Cancer Screening Programme. Gut. 2012 Jul;61(7):1050-7. doi: 10.1136/gutjnl-2011-300651. Epub 2011 Sep 22. PMID 21940723
- [Background] Lieberman D, Moravec M, Holub J, Michaels L, Eisen G. Polyp size and advanced histology in patients undergoing colonoscopy screening: implications for CT colonography. Gastroenterology. 2008 Oct;135(4):1100-5. doi: 10.1053/j.gastro.2008.06.083. Epub 2008 Jul 3. PMID 18691580
- [Background] Chen SC, Rex DK. Endoscopist can be more powerful than age and male gender in predicting adenoma detection at colonoscopy. Am J Gastroenterol. 2007 Apr;102(4):856-61. doi: 10.1111/j.1572-0241.2006.01054.x. Epub 2007 Jan 11. PMID 17222317
- [Background] Rex DK, Overhiser AJ, Chen SC, Cummings OW, Ulbright TM. Estimation of impact of American College of Radiology recommendations on CT colonography reporting for resection of high-risk adenoma findings. Am J Gastroenterol. 2009 Jan;104(1):149-53. doi: 10.1038/ajg.2008.35. PMID 19098863
- [Background] Butterly LF, Chase MP, Pohl H, Fiarman GS. Prevalence of clinically important histology in small adenomas. Clin Gastroenterol Hepatol. 2006 Mar;4(3):343-8. doi: 10.1016/j.cgh.2005.12.021. PMID 16527698
- [Background] Cairns S, Scholefield JH. Guidelines for colorectal cancer screening in high risk groups. Gut. 2002 Oct;51 Suppl 5(Suppl 5):V1-2. doi: 10.1136/gut.51.suppl_5.v1. PMID 12221029
- [Background] Levin B, Lieberman DA, McFarland B, Andrews KS, Brooks D, Bond J, Dash C, Giardiello FM, Glick S, Johnson D, Johnson CD, Levin TR, Pickhardt PJ, Rex DK, Smith RA, Thorson A, Winawer SJ; American Cancer Society Colorectal Cancer Advisory Group; US Multi-Society Task Force; American College of Radiology Colon Cancer Committee. Screening and surveillance for the early detection of colorectal cancer and adenomatous polyps, 2008: a joint guideline from the American Cancer Society, the US Multi-Society Task Force on Colorectal Cancer, and the American College of Radiology. Gastroenterology. 2008 May;134(5):1570-95. doi: 10.1053/j.gastro.2008.02.002. Epub 2008 Feb 8. PMID 18384785
- [Background] Lieberman DA, Weiss DG, Harford WV, Ahnen DJ, Provenzale D, Sontag SJ, Schnell TG, Chejfec G, Campbell DR, Kidao J, Bond JH, Nelson DB, Triadafilopoulos G, Ramirez FC, Collins JF, Johnston TK, McQuaid KR, Garewal H, Sampliner RE, Esquivel R, Robertson D. Five-year colon surveillance after screening colonoscopy. Gastroenterology. 2007 Oct;133(4):1077-85. doi: 10.1053/j.gastro.2007.07.006. PMID 17698067
- [Background] ASGE TECHNOLOGY COMMITTEE; Song LM, Adler DG, Conway JD, Diehl DL, Farraye FA, Kantsevoy SV, Kwon R, Mamula P, Rodriguez B, Shah RJ, Tierney WM. Narrow band imaging and multiband imaging. Gastrointest Endosc. 2008 Apr;67(4):581-9. doi: 10.1016/j.gie.2008.01.013. PMID 18374021
- [Background] Cohen J. Optical contrast endoscopy: is it ready for routine use? Gastroenterology. 2009 Jan;136(1):52-5. doi: 10.1053/j.gastro.2008.11.053. Epub 2008 Dec 6. No abstract available. PMID 19063888
- [Background] East JE, Suzuki N, Saunders BP. Comparison of magnified pit pattern interpretation with narrow band imaging versus chromoendoscopy for diminutive colonic polyps: a pilot study. Gastrointest Endosc. 2007 Aug;66(2):310-6. doi: 10.1016/j.gie.2007.02.026. PMID 17643705
- [Background] Konerding MA, Fait E, Gaumann A. 3D microvascular architecture of pre-cancerous lesions and invasive carcinomas of the colon. Br J Cancer. 2001 May 18;84(10):1354-62. doi: 10.1054/bjoc.2001.1809. PMID 11355947
- [Background] Sano Y, Ikematsu H, Fu KI, Emura F, Katagiri A, Horimatsu T, Kaneko K, Soetikno R, Yoshida S. Meshed capillary vessels by use of narrow-band imaging for differential diagnosis of small colorectal polyps. Gastrointest Endosc. 2009 Feb;69(2):278-83. doi: 10.1016/j.gie.2008.04.066. Epub 2008 Oct 25. PMID 18951131
- [Background] Hirata M, Tanaka S, Oka S, Kaneko I, Yoshida S, Yoshihara M, Chayama K. Evaluation of microvessels in colorectal tumors by narrow band imaging magnification. Gastrointest Endosc. 2007 Nov;66(5):945-52. doi: 10.1016/j.gie.2007.05.053. PMID 17963882
- [Background] Rogart JN, Jain D, Siddiqui UD, Oren T, Lim J, Jamidar P, Aslanian H. Narrow-band imaging without high magnification to differentiate polyps during real-time colonoscopy: improvement with experience. Gastrointest Endosc. 2008 Dec;68(6):1136-45. doi: 10.1016/j.gie.2008.04.035. Epub 2008 Aug 8. PMID 18691708
- [Background] Rastogi A, Pondugula K, Bansal A, Wani S, Keighley J, Sugar J, Callahan P, Sharma P. Recognition of surface mucosal and vascular patterns of colon polyps by using narrow-band imaging: interobserver and intraobserver agreement and prediction of polyp histology. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):716-22. doi: 10.1016/j.gie.2008.09.058. PMID 19251016
- [Background] East JE, Suzuki N, Bassett P, Stavrinidis M, Thomas HJ, Guenther T, Tekkis PP, Saunders BP. Narrow band imaging with magnification for the characterization of small and diminutive colonic polyps: pit pattern and vascular pattern intensity. Endoscopy. 2008 Oct;40(10):811-7. doi: 10.1055/s-2008-1077586. Epub 2008 Sep 30. PMID 18828077
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] Atkin WS, Saunders BP; British Society for Gastroenterology; Association of Coloproctology for Great Britain and Ireland. Surveillance guidelines after removal of colorectal adenomatous polyps. Gut. 2002 Oct;51 Suppl 5(Suppl 5):V6-9. doi: 10.1136/gut.51.suppl_5.v6. No abstract available. PMID 12221031
- [Background] Hassan C, Pickhardt PJ, Rex DK. A resect and discard strategy would improve cost-effectiveness of colorectal cancer screening. Clin Gastroenterol Hepatol. 2010 Oct;8(10):865-9, 869.e1-3. doi: 10.1016/j.cgh.2010.05.018. Epub 2010 Jun 1. PMID 20621680
- [Background] Ignjatovic A, Thomas-Gibson S, East JE, Haycock A, Bassett P, Bhandari P, Man R, Suzuki N, Saunders BP. Development and validation of a training module on the use of narrow-band imaging in differentiation of small adenomas from hyperplastic colorectal polyps. Gastrointest Endosc. 2011 Jan;73(1):128-33. doi: 10.1016/j.gie.2010.09.021. PMID 21184878
- [Background] World Health Organisation. World Health Organisation classification of tumours:pathology and genetics of tumours of the digestive system. Lyon: IARC press. 2000.
- [Background] NHS Bowel Cancer Screening Programme: Quality Assurance Guidelines for Colonoscopy. Andrew Chilton and Matt Rutter. March 2010. Available at: http://www.cancerscreening.nhs.uk/bowel/publications/nhsbcsp06.html
- [Derived] Rees CJ, Rajasekhar PT, Wilson A, Close H, Rutter MD, Saunders BP, East JE, Maier R, Moorghen M, Muhammad U, Hancock H, Jayaprakash A, MacDonald C, Ramadas A, Dhar A, Mason JM. Narrow band imaging optical diagnosis of small colorectal polyps in routine clinical practice: the Detect Inspect Characterise Resect and Discard 2 (DISCARD 2) study. Gut. 2017 May;66(5):887-895. doi: 10.1136/gutjnl-2015-310584. Epub 2016 Apr 19. PMID 27196576